CLINICAL TRIAL: NCT06002295
Title: A Comparative Analysis of 4% Chlorhexidine Versus Methylated Spirit as Prophylaxis of Omphalitis and Sepsis in Newborns
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Responsible Party: Principal Investigator, Ahmad Zunair Wasim, Resident Doctor, Sheikh Zayed Federal Postgraduate Medical Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZMC/IRB/Internal/MD/130/19
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Neonatal Sepsis; Omphalitis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Umbilical Cord Care with Chlorhexidine (Group A) (Experimental)
  Interventions: Drug: Chlorhexidine Topical Cream
- Umbilical Cord Care with Methylated Spirit (Group B) (Experimental)
  Interventions: Drug: Methylated Spirit

INTERVENTIONS:
Drug: Chlorhexidine Topical Cream — After approval from the hospital ethical committee, neonates fulfilling inclusion and exclusion criteria were selected. Written informed consent was obtained from the parents. Full instructions to avoid confounding variables like maintaining temperature and hygiene of newborn, frequent diaper change, avoidance of herbal tonics and cow milk; are given to mothers.
  In group "A" 4% chlorhexidine was applied generously over cord along with base of cord stump and surrounding skin thrice a day. In group "B" clean cotton swab dipped in methylated spirit was used to clean cord along with cord clamps and base thrice a day.
  Arms: Umbilical Cord Care with Chlorhexidine (Group A)
Drug: Methylated Spirit — After approval from the hospital ethical committee, neonates fulfilling inclusion and exclusion criteria were selected. Written informed consent was obtained from the parents. Full instructions to avoid confounding variables like maintaining temperature and hygiene of newborn, frequent diaper change, avoidance of herbal tonics and cow milk; are given to mothers.
  In group "A" 4% chlorhexidine was applied generously over cord along with base of cord stump and surrounding skin thrice a day. In group "B" clean cotton swab dipped in methylated spirit was used to clean cord along with cord clamps and base thrice a day.
  Arms: Umbilical Cord Care with Methylated Spirit (Group B)

SUMMARY:
Introduction: Neonatal sepsis in one of the leading cause of death in developing countries. Umbilical cord care is important as it may lead to infection. Topical treatment can help to reduce the chances of infection as well as increase the chances of early removal. In this regard methylated spirit and chlorhexidine are found to be effective.

Aims and Objectives: To compare the effectiveness of 4% chlorhexidine and methylated spirit in newborns for prevention of omphalitis and neonatal sepsis.

Materials and Methods: This randomized control trial was carried out in neonatal unit of Shaikh Zayed Hospital Lahore. After meeting the inclusion criteria, 300 neonates were enrolled. In group A 4% chlorhexidine was applied for cord care and in group B methylated spirit was used. Neonates were followed till 10th day of life. Careful examination was done for cord separation and for any signs of omphalitis or sepsis. If the neonate had no signs and symptoms of omphalitis and sepsis on 10th day of follow up then it was treatment success.

DETAILED DESCRIPTION:
Introduction:

Neonatal sepsis in one of the leading causes of death in neonates in developing countries. Infection of the umbilical cord often leads to infection in the blood. World Health Organization (WHO) recommends 4% chlorhexidine to prevent omphalitis and neonatal sepsis. In Pakistan the investigators use methylated spirit for prophylaxis of omphalitis as 4% chlorhexidine is not available and expensive to use. Some commercial gels containing 2% chlorhexidine is available, but these are not as effective as methylated spirit.

Chlorhexidine gel is an antiseptic agent with broad-spectrum bactericidal and bacteriostatic properties effective against gram-negative bacteria and fungi with rapid pathogen killing rates. Methylated spirit on the other hand is both bactericidal, mycobactericidal, fungicidal, and viricidal agent.

In Pakistan Staphylococcal aureus is common pathogen in umbilical discharge. Some low cost prevention therapy should be used. Methylated spirit is commonly used for cord care. A study was conducted to explore about cord care practices in African setting which showed that 73.2% respondents consider methylated spirit as most important agent for cord care.

Chlorhexidine is available in different concentrations for antiseptic purpose. Efficacy of all concentrations is comparable but 4% chlorhexidine concentration is more effective in inhibiting organism's flora as compared to 2% chlorhexidine. Since then, multiple studies were done to compare between methylated spirit and 4% chlorhexidine. Methylated spirit is equally safe where 4% chlorhexidine is unavailable.

In Pakistan 57% deaths occur in neonatal period. Pakistan has highest neonatal mortality rate of 42 per 1000 live births. In developing countries neonatal sepsis is aggravated by home deliveries, antibiotic resistance and less medical staff. The most important way to decrease mortality and morbidity due to infections is prevention at an early stage. According to a study conducted in Karachi, omphalitis is 217.4/1000 live births from which moderate-severe omphalitis is 170/1000 live births and associated with sepsis is 20.4/1000 live births. Various antiseptics used in neonatal intensive care units include chlorhexidine, alcohol, iodine, hexachlorophene & octenidine. Each agent having its own advantages and adverse effects. However best antiseptic is yet to be determined.

World Health Organization (WHO) recommends application for 4 percent chlorhexidine in high neonatal mortality area and methylated spirit for cord care while methylated spirit is commonly used agent for cord care. One study conducted shows that applying chlorhexidine on cord in neonatal intensive care unit decreases mortality rate and decreases time of separation of cord.

Methylated spirit and chlorhexidine both have comparable efficacy and can be used in areas of non-availability of chlorhexidine and whenever chlorhexidine is not safe to use as in very preterm neonates. In Pakistan there is no population based study published on this issue this study aimed to compare the effectiveness of methylated spirit and 4% chlorohexidine from prevention of omphalitis and neonatal sepsis. This study will help to establish the use of methylated spirit in prevention of omphalitis and neonatal sepsis at low price and easy availability.

Methodology:

It was a randomized controlled trial done at the Neonatology unit, Department of Pediatrics, Shaikh Zayed Hospital, Lahore. For a period of 12 months from September 2020 to September 2021 with the hypothesis that methylated spirit is equally effective as 4% chlorhexidine in preventing omphalitis and sepsis in neonate. 300 newborns were included by probability consecutive sampling in study with 150 newborns in each group with confidence interval of 95% and margin of error 5%. Sample size was calculated using Raosoft sample size calculator.

After approval from the hospital ethical committee, neonates fulfilling inclusion and exclusion criteria were selected. Written informed consent was obtained from the parents. Full instructions to avoid confounding variables like maintaining temperature and hygiene of newborn, frequent diaper change, avoidance of herbal tonics and cow milk were given to mothers.

In group "A" mothers were advised the topical application of 4% chlorhexidine generously over cord along with base of cord stump and surrounding skin thrice a day. In group "B" clean cotton swab dipped in methylated spirit was used to clean cord along with cord clamps and base thrice a day.

Neonates were followed till 10th day of life and careful examination was done for cord separation and any signs of omphalitis or sepsis. Primary outcome measure was omphalitis which was characterized by local inflamed cord. Secondary outcome measure was sepsis which was characterized by signs and symptoms such as fever, reluctance to feed, respiratory difficulty, irritability. Treatment success was labelled if there was no evidence of omphalitis or sepsis. If omphalitis or evidence of sepsis was present, the patient was treated as per hospital protocol. Data was collected according to proforma.

Statistical Analysis:

Data was entered in SPSS v.23.0 and was analyzed through it. The numeric variables like gestational age at birth and birth weight were presented as mean ± standard deviation, while the categorical variables like gender of the neonate, omphalitis and sepsis were presented as frequency (%). Both groups were compared for omphalitis and sepsis by using the chi-square (ﬡ²) test. P-value ≤ 0.05 was kept as significant. Data was stratified for gender of the neonate, gestational age at birth and birth weight to deal with the effect modifiers. Post-stratification, Chi-Square test was applied to compare both groups for omphalitis and sepsis in each strata. P-value ≤ 0.05 was kept as significant.

ELIGIBILITY:
Inclusion Criteria:

* Term neonates of either gender born via cesarean section or spontaneous vaginal delivery at Shaikh Zayed Hospital after taking informed consent of parents.
* Antiseptic agent started from 1st day of life & up to 10 days continued without missing dose

Exclusion Criteria:

* Newborns with congenital defects or cord anomalies.
* Laboratory or clinical evidence of sepsis.
* Preterm newborns
* Newborns having very low birth weight <1.5 kg
* Any evidence of asphyxia during birth.

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with Omphalitis | 10 days
  Inflammation of the navel in newborn babies as assessed by redness and swelling of the area.

SECONDARY OUTCOMES:
Number of participants with Neonatal Sepsis | 10 days
  It refers to an infection involving bloodstream in newborn infants less than 28 days old as assessed by following parameters: fever >38.5 °, heart rate >2SD for age, respiratory rate >2SD for age, irritability, lethargic, cyanosis, poor perfusion, feeding difficulty, urine output <0.5ml/kg/hr.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh Zayed Federal Postgraduate Medical Institute, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No